CLINICAL TRIAL: NCT05082922
Title: Implementation of a Transdiagnostic Emotion-focused Treatment for Comorbid Emotional Problems and Chronic Pain in Clinical Care. A Sequential Replicated and Randomized Single Case Experimental Design (SCED).
Brief Title: Implementation of the Hybrid Treatment in Clinical Care. A SCED.
Acronym: hybrid-sced
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HYBRID2.0
Record Dates: First submitted 2021-10-01; First posted 2021-10-19 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Emotional Problem; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: This study employs a sequential single-case experimental AB design with randomized waiting period lengths (4, 5 or 6 weeks). Included in the design is also standardized pre-post and follow up measurement allowing for single group analysis of change. In addition, we collect qualitative data from patients, practitioners and clinical managers, detailing how the treatment and its implementation are experienced.
Who Masked: Outcomes Assessor
Masking Description: Data is collected using a secure digital platform. Outcome assessors will be blinded to baseline length allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No treatment waiting period (No Intervention): Participants are randomized to a 4, 5, or 6 week waiting period. Weekly measurements are collected throughout this period.
- Hybrid treatment (Experimental): Hybrid treatment. Weekly measurements are collected throughout treatment.
  Interventions: Behavioral: Hybrid treatment

INTERVENTIONS:
Behavioral: Hybrid treatment — Transdiagnostic emotion-focused treatment provided by a psychologist with, when needed, support of a medical doctor (ensuring adherence to medical guidelines) and a physiotherapist (providing assessment and treatment support in exposure for physical activities). Depending on the length of the waiting period (randomly assigned to be either 4, 5 or 6 weeks), the treatment period varies between 14-16 weeks and contains 10-15 sessions.
  Arms: Hybrid treatment

SUMMARY:
In society today, mental health problems, specifically stress-, anxiety- and depressive disorders, are a primary cause of long-term sick leave, leading to significant societal costs and suffering. One important issue hindering implementation of successful treatments is that there is a marked co-occurrence between these problems and somatic health problems, such as different types of pain. An important key to solving this problem is to develop a more integrated conceptualization of, and treatment model for, these patients' health problems. Specifically, one way to understand the co-occurrence between mental and somatic health problems is offered by the 'transdiagnostic' perspective. The aim of this project is to implement and evaluate the effectiveness of a transdiagnostic emotion-focused treatment protocol in clinical context. The treatment addresses comorbid mental (stress, anxiety- and depressive) and somatic health (pain) problems and targets core emotion regulation processes that are hypothesized to maintain and exacerbate these problems.

ELIGIBILITY:
Inclusion Criteria:

* > 11 points on the anxiety or depression subscale, Hospital Anxiety and Depression scale
* somatic health problems (pain > 3 months) with functional impairment (>3 on question 2 of the Multidimensional Pain Inventory, MPI, OR > 20 points on question 21-24 of the Örebro Musculoskeletal Pain Questionnaire, ÖMPQ)

Exclusion Criteria:

* severe psychiatric problems requiring immediate other treatment
* current psychological treatment
* recently started psychopharmacological treatment for anxiety or depression (<3 months prior to planned treatment)
* insufficient mastery of the Swedish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Generalised Anxiety Disorder (GAD-7) change | repeated weekly through phase A (randomly assigned to be 4, 5 or 6 weeks) and treatment phase B (14 to 16 weeks). Total time frame of assessment is 20 weeks.
  change in self rated anxiety. Scale range 0-27 (higher values worse outcome)
Patient Health Questionnaire (PHQ-9) change | repeated weekly through phase A (randomly assigned to be 4, 5 or 6 weeks) and treatment phase B (14 to 16 weeks). Total time frame of assessment is 20 weeks.
  change in self rated depression. Scale range 0-27 (higher values worse outcome)
Pain change | repeated weekly through phase A (randomly assigned to be 4, 5 or 6 weeks) and treatment phase B (14 to 16 weeks). Total time frame of assessment is 20 weeks.
  change in pain intensity (scale 0-6) and interference. Scale range 0-6 (higher values worse outcome)
Pain coping change | repeated weekly through phase A (randomly assigned to be 4, 5 or 6 weeks) and treatment phase B (14 to 16 weeks). Total time frame of assessment is 20 weeks.
  change in pain worry (scale 0-6) and avoidance (scale range 0-8) (higher values worse outcome)
Symptom Catastrophizing Scale (SCS) change | Baseline, 5 months and 11 months as well as repeated weekly through phase A (randomly assigned to be 4, 5 or 6 weeks) and treatment phase B (14 to 16 weeks). Total time frame of assessment is 20 weeks.
  Change in catastrophic interpretation of symptoms. Scale range 0-14 (higher values worse outcome)

SECONDARY OUTCOMES:
Multidimensional Pain Inventory (MPI) change | Baseline, 5 months and 11 months
  change in pain intensity and interference. Subscale pain intensity range 0-12, subscale pain interference range 0-66 (for both sub scales higher values worse outcome)
Montgomery Åsberg Depression Rating Scale (MADRS) change | Baseline, 5 months and 11 months
  change in self rated depression. Scale range 0-60 (higher values worse outcome)
Difficulties in Emotion Regulation Scale (DERS-16) change | Baseline, 5 months and 11 months
  change in emotion regulation abilities. Scale range 16-80 (higher values worse outcome)
Psychological Inflexibility in Pain Scale (PIPS) change | Baseline, 5 months and 11 months
  change in avoidance of pain (scale range 8-56) and fusion with pain thoughts (scale range 4-28) (higher values worse outcomes)
Work limitation questionnaire-16 change | Baseline, 5 months and 11 months
  change in thoughts and adaptations regarding work limitations due to symptoms. Scale range 16-80 (higher values worse outcomes).
Insomnia Sleep Inventory (ISI) change | Baseline, 5 months and 11 months
  change in insomnia. Scale range 0-28 (higher values worse outcome)
EQ5-D change | Baseline, 5 months and 11 months
  Health related quality of life. Scale range 0-100 (higher values worse outcome)
Mini international neuropsychiatric interview (MINI) | Baseline, 5 months
  Diagnostic screening interview-DSM-V

OTHER OUTCOMES:
adverse effects | 5 months
  adverse treatment effects
Treatment satisfaction questionnaire | 5 months
  self reported satisfaction with treatment
sick leave and medication use | Baseline, 5 months and 11 months
  self reported and national register derived information of sickleave and medication use. related to symptoms
experience of treatment | 5 months
  semi structured interviews probing qualitative aspects of the treatment experience, and the experience of implementation of patients, treating practitioners and clinical managers

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Health and Medical Psychology, Örebro, Sweden